CLINICAL TRIAL: NCT01747928
Title: A Representative Users Study Of The Operating Characteristics Of The Caverject Delivery System
Brief Title: Users Study Of The Caverject Delivery System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None
Other Study IDs: A6711036
Record Dates: First submitted 2012-11-20; First posted 2012-12-12 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: usability study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental)
  Interventions: Other: dual-chamber syringe

INTERVENTIONS:
Other: dual-chamber syringe — dual-chamber syringe for mock injection

SUMMARY:
Usability testing of the dual-chambered syringe in conjunction with the proposed patient instructions for use.

DETAILED DESCRIPTION:
Usability testing of the dual-chambered syringe in conjunction with the proposed patient instructions for use

ELIGIBILITY:
Inclusion Criteria:

* Healthy males

Exclusion Criteria:

* Inability to read English;
* physical limitations preventing participant from operating the syringe

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6711036&StudyName=Users%20Study%20Of%20The%20Caverject%20Delivery%20System%0A

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 50 participants were screened, among whom 2 did not meet entrance criteria. The remaining 48 participants did and were randomized to study treatment.
Groups:
- Caverject 10 mcg Device - 2.5 mcg Dose Setting: Participants used the 10 microgram (mcg) Caverject Impulse Dual Chamber Delivery System to expel alprostadil 2.5 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
- Caverject 10 mcg Device - 5 mcg Dose Setting: Participants used the 10 mcg Caverject Impulse Dual Chamber Delivery System to expel alprostadil 5.0 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
- Caverject 10 mcg Device - 7.5 mcg Dose Setting: Participants used the 10 mcg Caverject Impulse Dual Chamber Delivery System to expel alprostadil 7.5 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
- Caverject 10 mcg Device - 10 mcg Dose Setting: Participants used the 10 mcg Caverject Impulse Dual Chamber Delivery System to expel alprostadil 10 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
- Caverject 20 mcg Device - 5 mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Dual Chamber Delivery System to expel alprostadil 5.0 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
- Caverject 20 mcg Device - 10 mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Dual Chamber Delivery System to expel alprostadil 10 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
- Caverject 20 mcg Device - 15 mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Dual Chamber Delivery System to expel alprostadil 15 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
- Caverject 20 mcg Device - 20 mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Dual Chamber Delivery System to expel alprostadil 20 mcg into a receptacle (rubber injection trainer). Participants did not receive study medication.
Period: Overall Study
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Started | 6 (Participants initiated the attempt to perform the injection task.) | 6 (Participants initiated the attempt to perform the injection task.) | 6 (Participants initiated the attempt to perform the injection task.) | 6 (Participants initiated the attempt to perform the injection task.) | 6 (Participants initiated the attempt to perform the injection task.) | 6 (Participants initiated the attempt to perform the injection task.) | 6 (Participants initiated the attempt to perform the injection task.) | 6 (Participants initiated the attempt to perform the injection task.)
Completed | 6 (Participants carried on assessment to a point where Observer could determine success/failure.) | 6 (Participants carried on assessment to a point where Observer could determine success/failure.) | 6 (Participants carried on assessment to a point where Observer could determine success/failure.) | 6 (Participants carried on assessment to a point where Observer could determine success/failure.) | 6 (Participants carried on assessment to a point where Observer could determine success/failure.) | 6 (Participants carried on assessment to a point where Observer could determine success/failure.) | 6 (Participants carried on assessment to a point where Observer could determine success/failure.) | 6 (Participants carried on assessment to a point where Observer could determine success/failure.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (9.1) | 52.7 (10.0) | 51.3 (9.0) | 53.5 (9.0) | 63.0 (2.5) | 55.3 (4.8) | 57.8 (6.8) | 51.8 (5.6) | 54.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Delivery System Success Rate (DSSR)
Description: DSSR was defined as percentage of participants who were able to successfully expel the selected dose from the Caverject Impulse Dual Chamber Delivery System when relying on the modified Instructions for Use (IFU). The process was considered successful if the attempt was observed and documented by study personnel AND the participant didn't receive any operational/"hands on" demonstration on how to operate the plunger from study personnel AND after performing all preparatory steps, the participant was able to expel the dose to the selected plunger stop-point without any unexpected interruption.
Time Frame: Day 1
Population: The full analysis set (FAS) consisted of all protocol defined valid attempts to perform the study procedure as documented in the Observer Assessment Tool (OAT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: All participants who delivered a predefined dose and volume of alprostadil (prostaglandin E1 [PGE1], Caverject) into a receptacle, using the assigned Caverject Impulse Dual Chamber Delivery System. Participants did not receive study medication and were monitored during the handling of the Caverject Impulse Dual Chamber Delivery System.
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting | All Participants
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
percentage of participants | 66.67 [NA to NA] — Confidence interval (CI) only calculated for all combined participants. | 66.67 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 83.33 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 89.58 [79.34 to 100.0]

2. Post Hoc Outcome: DSSR Based on the Primary Objective
Description: This post-hoc DSSR was calculated in order to provide a DSSR that recognized as a "failure" only those participants who were unable to successfully complete the overall injection task, regardless of whether they met with difficulties at any step.
Time Frame: Day 1
Population: The FAS consisted of all protocol defined valid attempts to perform the study procedure as documented in the OAT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting | All Participants
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
percentage of participants | 83.33 [NA to NA] — CI only calculated for all combined participants. | 83.33 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 83.33 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 100.00 [NA to NA] — CI only calculated for all combined participants. | 93.75 [84.63 to 100.0]

3. Secondary Outcome: Number of Participants With Categorical Responses to the Participant Assessment Tool (PAT): Instructions Provided Were Useful?
Description: Participant responses were reported as follows: Very Useful, Somewhat Useful, Not Very Useful, Not Useful At All.
Time Frame: Day 1
Population: The FAS consisted of all protocol defined valid attempts to perform the study procedure as documented in the OAT.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Very useful | 5 | 5 | 6 | 5 | 6 | 5 | 5 | 6
  Somewhat useful | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Not very useful | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Not useful at all | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing answer | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Categorical Responses to the PAT: Instructions Provided Were Clear?
Description: Participant responses were reported as follows: Very clear, Somewhat clear, Not very clear, Not clear at all.
Time Frame: Day 1
Population: The FAS consisted of all protocol defined valid attempts to perform the study procedure as documented in the OAT.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Very clear | 5 | 4 | 6 | 6 | 6 | 5 | 5 | 5
  Somewhat clear | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1
  Not very clear | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not clear at all | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing answer | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Categorical Responses to the PAT: Most Difficult Step?
Description: Participant responses were reported as follows: No steps really difficult, Attaching needle, Mixing the solution, Getting the air out of syringe, Setting the dose, Pushing plunger, Other.
Time Frame: Day 1
Population: The FAS consisted of all protocol defined valid attempts to perform the study procedure as documented in the OAT.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  No steps really difficult | 5 | 3 | 4 | 5 | 6 | 4 | 5 | 5
  Attaching needle | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 0
  Mixing the solution | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Getting the air out of syringe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Setting the dose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Pushing plunger | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Missing answer | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Categorical Responses to the PAT: Syringe Easy to Use?
Description: Participant responses were reported as follows: Very easy, Somewhat easy, Somewhat difficult, Very difficult.
Time Frame: Day 1
Population: The FAS consisted of all protocol defined valid attempts to perform the study procedure as documented in the OAT.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Very easy | 4 | 3 | 5 | 6 | 6 | 5 | 6 | 6
  Somewhat easy | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0
  Somewhat difficult | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Very difficult | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing answer | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Providing Responses to Any Question on the PAT
Description: Number of participants providing responses on questions in the PAT. Questions were as follows: What step did you stop? Why?; Instructions provided were useful?; Instructions provided were clear?; Most difficult step?; Syringe easy to use?
Time Frame: Day 1
Population: The FAS consisted of all protocol defined valid attempts to perform the study procedure as documented in the OAT.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  What step did you stop? Why? | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Instructions provided were useful? | 5 | 6 | 6 | 6 | 6 | 6 | 5 | 6
  Instructions provided were clear? | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Most difficult step? | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Syringe easy to use? | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6

8. Secondary Outcome: Time Required to Perform Segments 1 to 5
Description: Steps involved while using the Caverject Impulse Delivery System were categorized into segments: Segment 1 (Assembly While Using the Caverject Impulse Delivery System), Segment 2 (Mixing the Solution), Segment 3 (De-aerating the Syring While Using the Caverject Impulse Delivery System), Segment 4 (Setting the Dose) and Segment 5 (Performing the Injection While Using the Caverject Impulse Delivery System).
Time Frame: Day 1
Population: The FAS consisted of all protocol defined valid attempts to perform the study procedure as documented in the OAT. n=number of participants analyzed for that segment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
seconds
  Segment 1 (n = 6, 6, 6, 6, 6, 6, 6, 6) | 148.8 (37.20) | 189.3 (140.13) | 176.0 (72.92) | 194.3 (107.53) | 246.5 (131.85) | 168.2 (82.76) | 142.3 (105.78) | 144.5 (23.35)
  Segment 2 (n = 5, 6, 6, 6, 6, 5, 6, 6) | 47.2 (21.53) | 73.0 (63.11) | 42.3 (14.19) | 53.8 (30.73) | 53.8 (21.68) | 50.2 (35.90) | 64.2 (50.03) | 39.5 (13.92)
  Segment 3 (n = 5, 6, 6, 6, 6, 5, 6, 6) | 49.2 (15.69) | 60.2 (40.41) | 71.8 (22.69) | 79.5 (89.17) | 55.8 (32.03) | 42.6 (5.86) | 43.2 (22.13) | 63.3 (24.82)
  Segment 4 (n = 5, 5, 6, 6, 6, 5, 6, 6) | 34.4 (29.55) | 37.4 (59.77) | 29.0 (23.08) | 30.0 (26.71) | 20.0 (13.07) | 8.4 (6.31) | 31.7 (24.20) | 35.7 (16.50)
  Segment 5 (n = 5, 5, 6, 6, 6, 5, 6, 6) | 30.4 (17.04) | 38.8 (53.64) | 30.3 (17.77) | 19.2 (11.96) | 30.8 (15.25) | 17.4 (13.24) | 27.3 (20.38) | 30.8 (17.51)

9. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q1
Description: OAT, Q1: Participant assembled the components correctly. Observer responses were reported as follows: Yes, No. A "No" answer indicated failure according to the OAT. Q1 and Q2 made up Segment 1: Assembly of Components.
Time Frame: Day 1
Population: FAS: all protocol defined valid attempts to perform the study procedures as documented in the OAT. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per OAT) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q2
Description: OAT, Q2: Evidence of mechanical malfunction or defect for Segment 1. Observer responses were reported as follows: Yes, No. Q1 and Q2 made up Segment 1: Assembly of Components.
Time Frame: Day 1
Population: FAS: all protocol defined valid attempts to perform the study procedures as documented in the OAT. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination. 1 participant in the 10 mcg device-2.5 mcg dose was excluded as failure at Q1 did not involve mechanical failure or defect.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Excluded from Q2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Whom the Observer Had Categorical Responses to in the OAT: Q3
Description: OAT, Q3: Participant performed mixing step correctly. Observer responses were reported as follows: Yes, No. A "No" response indicated failure according to the OAT. Q3 to Q5 made up Segment 2: Mixing the Solution.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination. 1 participant each in the 10 mcg device-2.5 mcg dose and the 20 mcg device-10 mcg dose were excluded as they failed in Segment 1 and did not proceed to Segment 2. These 2 participants are counted in the "did not participate" category.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per OAT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

12. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q4
Description: OAT, Q4: Participant positioned piston correctly. Observer responses were reported as follows: Yes, No. A "No" response indicated failure according to the SAP. Q3 to Q5 made up Segment 2: Mixing the Solution.
Time Frame: Day 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per SAP) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

13. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q5
Description: OAT, Q5: Evidence of mechanical malfunction/defect for Segment 2. Observer responses were reported as follows: Yes, No. Q3 to Q5 made up Segment 2: Mixing the Solution.
Time Frame: Day 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 6
  Did not participate | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q6
Description: OAT, Q6: De-aeration step performed successfully. Observer responses were reported as follows: Yes, No. A "No" response indicated failure according to the OAT. Q6 to Q8 made up Segment 3: De-aeration of the Syringe.
Time Frame: Day 1
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per OAT) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

15. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q7
Description: OAT, Q7: Participant depressed the plunger correctly to de-aerate the syringe. Observer responses were reported as follows: Yes, No. A "No" response indicated failure according to the SAP. Q6 to Q8 made up Segment 3: De-aeration of the Syringe.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per SAP) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

16. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q8
Description: OAT, Q8: Evidence of mechanical malfunction/defect for Segment 3. Observer responses were reported as follows: Yes, No. Q6 to Q8 made up Segment 3: De-aeration of the Syringe.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

17. Secondary Outcome: Number of Participants Whom the Observer Had Categorical Responses to in the OAT: Q9
Description: OAT, Q9: Participant was able to set a dose (any dose) for delivery. Observer responses were reported as follows: Yes, No. A "No" response indicated failure according to the OAT. Q9 and Q10 made up Segment 4: Setting the Dose.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per OAT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

18. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q10
Description: OAT, Q10: Evidence of mechanical malfunction/defect for Segment 4. Observer responses were reported as follows: Yes, No. Q9 and Q10 made up Segment 4: Setting the Dose.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

19. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q11
Description: OAT, Q11: Participant successfully set the correct dose (as assigned). Observer responses were reported as follows: Yes, No. A "No" response indicated failure according to the OAT. Q11 to Q17 made up Segment 5: Performing the Simulated Injection.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per OAT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

20. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q12
Description: OAT, Q12: Participant successfully expelled the dose into the target. Observer responses were reported as follows: Yes, No. A "No" response indicated failure according to the OAT. Q11 to Q17 made up Segment 5: Performing the Simulated Injection.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  No (FAIL per OAT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

21. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q13
Description: OAT, Q13: Was there any difficulty/obstruction encountered in expelling dose? Observer responses were reported as follows: Yes, No. A "Yes" response indicated failure according to the SAP. Q11 to Q17 made up Segment 5: Performing the Simulated Injection.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes (FAIL per SAP) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  No | 4 | 4 | 6 | 6 | 6 | 5 | 6 | 6
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

22. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q14b
Description: OAT, Q14b: Participant successfully expelled/injected the assigned dose (per Dose Card). Observer responses were reported as follows: Yes, No. Q11 to Q17 made up Segment 5: Performing the Simulated Injection.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  No | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

23. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q16
Description: OAT, Q16: Evidence of mechanical malfunction/defect. Observer responses were reported as follows: Yes, No. Q11 to Q17 made up Segment 5: Performing the Simulated Injection.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

24. Secondary Outcome: Number of Participants Which the Observer Had Categorical Responses to in the OAT: Q17
Description: OAT, Q17: Participant understood reason excess liquid was present after a partial-dose injection. Observer responses were reported as follows: Yes, No. Q11 to Q17 made up Segment 5: Performing the Simulated Injection.
Time Frame: Day 1
Population: FAS. All 48 participants were included in the FAS. Each participant tested 1 device/dose combination. All participants in the 10 mcg device-10 mcg dose and 20 mcg device-20 mcg dose (total 12 participants) are stated as "not applicable" as they tested the full dose.
Measure: Number; unit: participants
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Yes | 5 | 5 | 6 | 0 | 6 | 5 | 6 | 0
  No | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Did not participate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Not applicable (tested full dose) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 6

ADVERSE EVENTS:
Arm/Group | Caverject 10 mcg Device - 2.5 mcg Dose Setting | Caverject 10 mcg Device - 5 mcg Dose Setting | Caverject 10 mcg Device - 7.5 mcg Dose Setting | Caverject 10 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 5 mcg Dose Setting | Caverject 20 mcg Device - 10 mcg Dose Setting | Caverject 20 mcg Device - 15 mcg Dose Setting | Caverject 20 mcg Device - 20 mcg Dose Setting
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
For outcome measure 7, the endpoint was originally the comments provided as part of the PAT. As clinicaltrials.gov do not support textual results, the number of participants who provided comments to any questions on the PAT are reported instead.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.